CLINICAL TRIAL: NCT03665818
Title: The Influence of Mandibular Advancement Device Treating OSAHS on Primary Prevention of Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Zhao, Director of the Department of Stomatology，Xuanwu Hospital, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA-Z2015-06
Record Dates: First submitted 2018-07-18; First posted 2018-09-11 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Sleep Apnea Syndromes; Atherosclerosis; Carotid Plaque
MeSH Terms: conditions — Sleep Apnea Syndromes; Atherosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral appliance intervention (Experimental)
  Interventions: Device: oral appliance treatment
- Without oral appliance intervention (No Intervention)

INTERVENTIONS:
Device: oral appliance treatment — mandibular advancement device to enlarge pharyngeal airway space to get rid of apnea and hypopnea events
  Arms: Oral appliance intervention

SUMMARY:
1. The purpose of this study is to detect the differences of carotid atherosclerosis severity between patients with or without OSAHS(Obstructive Sleep Apnea and Hypopnea Syndrome) in a cross-sectional study in a large sample.
2. Then a longitudinal control study is conducted to observe the progress of the carotid atherosclerosis by vascular ultrasonography and the occurrence of cerebrovascular events after the intervention of the oral appliance for treating OSAHS，and finally explore the feasibility of using oral appliance to treat OSAHS in primary prevention of ischemic stroke.

DETAILED DESCRIPTION:
1. the relevance of OSAHS and carotid atherosclerosis Patients are distributed questionnaire and recruited from neurology clinic，vascular ultrasonography clinic of Xuanwu Hospital if they match the inclusion criteria. After initial screening, carotid atherosclerosis patients with skeptical OSAHS are sent to sleep center for polysomnography examination to determine the severity of OSAHS. At least 50 patients for mild, moderate, severe OSAHS each are recruited for OSAHS Group. At least 100 patients without snoring from questionnaire and without OSAHS after PSG screening are recruited for non OSAHS Group. Vascular ultrasonography examination for carotid are done for the two groups. Data of carotid vascular plaque from two groups are collected. Statistics are done to detect differences of carotid atherosclerosis severity between patients with and without OSAHS, also the severity of OSAHS.
2. the relevance of the progress of carotid atherosclerosis and oral appliances intervention for treating OSAHS All carotid atherosclerosis patients with OSAHS are from patients of the first study. If they consent the treatment of oral appliances, they are recruited into this second study. At least 100 patients are recruited. They are divided into 2 groups by randomized block design by Evidence-based Medicine Center of Xuanwu Hospital. One group is oral appliance intervention group, the other group is no intervention group. The intervention group patients accept oral appliance treatment, and no intervention group patients do not accept OSAHS treatment. The two groups both accept anti-hypertension treatment or anti-diabetes treatment, or anti-hyperlipidemia treatment according to their own situation in neurology clinic.

At timepoint of initial time, one month after oral appliance treatment, one and a half year after oral appliance treatment, the intervention group should accept PSG(Polysomnography) examination to monitor the treatment of OSAHS.

At timepoint of initial time, one month after oral appliance treatment, one and a half year after oral appliance treatment, the two groups should accept breath holding test to monitor the cerebral vascular reserve.

At timepoint of initial time, one and a half year after oral appliance treatment, the two groups should accept carotid vascular ultrasonography examination to monitor the progress of carotid atherosclerosis.

Cerebrovascular events and death are recorded from initial time. Statistics are done to detect the influence of treatment of OSAHS on carotid atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with atherosclerosis by vascular ultrasonography
* diagnosed with OSAHS by polysomnography

Exclusion Criteria:

* patients who have stroke already
* patients who can not wear oral appliances according to experiment requirements
* patients who have bad periodontal condition or teeth number less than 20

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07-09 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
apnea hypopnea events 0 in Times | initial time when patients are recruited
  apnea and hypopnea times per hour
apnea hypopnea events 1 in Times | one month after oral appliance treatment
  apnea and hypopnea times per hour
apnea hypopnea events 2 in Times | one and a half years after oral appliance treatment
  apnea and hypopnea times per hour
longest apnea time 0 in Seconds | initial time when patients are recruited
  longest apnea or hypopnea time
longest apnea time 1 in Seconds | one month after oral appliance treatment
  longest apnea or hypopnea time
longest apnea time 2 in Seconds | one and a half years after oral appliance treatment
  longest apnea or hypopnea time
Blood oxygen saturation less than 90% of the total monitoring time percentage 0 in percentage | initial time when patients are recruited
  Blood oxygen saturation less than 90% of the total monitoring time percentage
Blood oxygen saturation less than 90% of the total monitoring time percentage 1 in percentage | one month after oral appliance treatment
  Blood oxygen saturation less than 90% of the total monitoring time percentage
Blood oxygen saturation less than 90% of the total monitoring time percentage 2 in percentage | one and a half years after oral appliance treatment
  Blood oxygen saturation less than 90% of the total monitoring time percentage
lowest Oxygen Saturation 0 in percentage | initial time when patients are recruited
  blood lowest oxygen saturation during the whole night
lowest Oxygen Saturation 1 in percentage | one month after oral appliance treatment
  blood lowest oxygen saturation during the whole night
lowest Oxygen Saturation 2 in percentage | one and a half years after oral appliance treatment
  blood lowest oxygen saturation during the whole night
atherosclerosis plaque thickness 0 in common carotid artery in milimetre | initial time when patients are recruited
  atherosclerosis plaque thickness is distance from the most convex point of plaque to carotid media
atherosclerosis plaque thickness 1 in common carotid artery in milimetre | one and a half years after oral appliance treatment
  atherosclerosis plaque thickness is distance from the most convex point of plaque to carotid media
atherosclerosis plaque length 0 in common carotid artery in milimetre | initial time when patients are recruited
  atherosclerosis plaque length is distance from the beginning to the end of a separate plaque
atherosclerosis plaque length 1 in common carotid artery in milimetre | one and a half years after oral appliance treatment
  atherosclerosis plaque length is distance from the beginning to the end of a separate plaqu
atherosclerosis plaque thickness 0 in internal carotid artery in milimetre | initial time when patients are recruited
  atherosclerosis plaque thickness is distance from the most convex point of plaque to carotid media
atherosclerosis plaque thickness 1 in internal carotid artery in milimetre | one and a half years after oral appliance treatment
  atherosclerosis plaque thickness is distance from the most convex point of plaque to carotid media
atherosclerosis plaque thickness 0 in carotid bulb in milimetre | initial time when patients are recruited
  atherosclerosis plaque thickness is distance from the most convex point of plaque to carotid media
atherosclerosis plaque thickness 1 in carotid bulb in milimetre | one and a half years after oral appliance treatment
  atherosclerosis plaque thickness is distance from the most convex point of plaque to carotid media
atherosclerosis plaque length 0 in internal carotid artery in milimetre | initial time when patients are recruited
  atherosclerosis plaque length is distance from the beginning to the end of a separate plaque
atherosclerosis plaque length 1 in internal carotid artery in milimetre | one and a half years after oral appliance treatment
  atherosclerosis plaque length is distance from the beginning to the end of a separate plaque
atherosclerosis plaque length 0 in carotid bolb in milimetre | initial time when patients are recruited
  atherosclerosis plaque length is distance from the beginning to the end of a separate plaque
atherosclerosis plaque length 1 in carotid bolb in milimetre | one and a half years after oral appliance treatment
  atherosclerosis plaque length is distance from the beginning to the end of a separate plaque
breath holding index 0 in percentage/seconds | initial time when patients are recruited
  breath holding index = (v2-v1)/v2*100/t. v2 is average velocity of middle cerebral artery after breath holding, v1 is average velocity of middle cerebral artery before breath holding, t is time for breath holding.
breath holding index 0 in percentage/seconds | one and a half years after oral appliance treatment
  breath holding index = (v2-v1)/v2*100/t. v2 is average velocity of middle cerebral artery after breath holding, v1 is average velocity of middle cerebral artery before breath holding, t is time for breath holding.
End systolic velocity of common carotid artery 0 in cm/s | initial time when patients are recruited
  the velocity of common carotid artery at the end of systolic period
End systolic velocity of common carotid artery 1 in cm/s | one and a half years after oral appliance treatment
  the velocity of common carotid artery at the end of systolic period
End systolic velocity of internal carotid artery 0 in cm/s | initial time when patients are recruited
  the velocity of internal carotid artery at the end of systolic period
End systolic velocity of internal carotid artery 1 in cm/s | one and a half years after oral appliance treatment
  the velocity of internal carotid artery at the end of systolic period
End systolic velocity of carotid bulb 0 in cm/s | initial time when patients are recruited
  the velocity of carotid bulb at the end of systolic period
End systolic velocity of carotid bulb 1 in cm/s | one and a half years after oral appliance treatment
  the velocity of carotid bulb at the end of systolic period
end diastolic velocity of common carotid artery 0 in cm/s | initial time when patients are recruited
  the velocity of common carotid artery at the end of diastolic period
end diastolic velocity of common carotid artery 1 in cm/s | one and a half years after oral appliance treatment
  the velocity of common carotid artery at the end of diastolic period
end diastolic velocity of internal carotid artery 0 in cm/s | initial time when patients are recruited
  the velocity of internal carotid artery at the end of diastolic period
end diastolic velocity of internal carotid artery 1 in cm/s | one and a half years after oral appliance treatment
  the velocity of internal carotid artery at the end of diastolic period
end diastolic velocity of carotid bulb 0 in cm/s | initial time when patients are recruited
  the velocity of carotid bulb at the end of diastolic period
end diastolic velocity of carotid bulb 1 in cm/s | one and a half years after oral appliance treatment
  the velocity of carotid bulb at the end of diastolic period

REFERENCES:
- [Derived] Qin L, Li N, Tong J, Hao Z, Wang L, Zhao Y. Impact of mandibular advancement device therapy on cerebrovascular reactivity in patients with carotid atherosclerosis combined with OSAHS. Sleep Breath. 2021 Sep;25(3):1543-1552. doi: 10.1007/s11325-020-02230-x. Epub 2021 Jan 7. PMID 33415656
- [Derived] Hao Z, Qin L, Tong J, Li N, Zhai Y, Zhao Y. The differences of carotid atherosclerosis among non-OSAHS and OSAHS patients of different severities: a cross-sectional study. Sleep Breath. 2021 Jun;25(2):639-648. doi: 10.1007/s11325-020-02145-7. Epub 2020 Jul 27. PMID 32720016